CLINICAL TRIAL: NCT00021775
Title: HIV Prevention Preparedness Study
Brief Title: HIV Prevention Preparedness Study in Russia, China, and India
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HPTN 033; 10611 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2001-08-04; First posted 2001-08-31 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: Risk Factors; Incidence; Patient Selection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to set up a system for doing research on HIV prevention in various parts of the world.

In order to plan large, long-term studies on the prevention of HIV in different areas of the world, it is necessary to get certain information first. It is important to know about the rate of HIV infection and how to get people to enroll for any future studies. This study will be done at 4 study locations.

DETAILED DESCRIPTION:
In order to realistically plan for future Phase III studies on HIV prevention, information must be obtained to characterize study population parameters at HTPN sites. Very different study designs may be required depending on these parameters, such as the ability of HPTN research centers to recruit study participants and the rate of HIV incidence observed in study populations. This study will be conducted at 4 HPTN sites to establish the necessary research knowledge and infrastructure.

This study enrolls participants from St. Petersburg, Russia; Xinjiang and Guangxi, China; and Chennai, India who are at high risk for HIV infection due to sexual and/or drug use behaviors. Participants who meet the screening criteria then complete an HIV risk assessment interview, receive HIV pre-test and risk reduction counseling, and undergo phlebotomy for HIV antibody testing. Participants who test positive are referred to available services and studies. Those who test HIV-negative and meet eligibility criteria are enrolled and maintained in follow-up over the next 12 months. Participants complete "locator contacts" at Months 3 and 9 and have follow-up visits at Months 6 and 12 for similar tests as performed at entry. In a substudy of this trial in China, participants will be interviewed about their drug use, social networks, needs, and perceptions about HIV/AIDS. These results will be used by HPTN to design more culturally sensitive and appropriate trials in the future.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are 16 (Saint Petersburg) or 18 (Xinjiang, Guangxi, and Chennai) years of age or older.
* Are HIV sero-negative.
* Are available for 12 months of study participation.
* Have written consent of parent or legal guardian if under age.
* Are able and willing to provide information on where they can be located or contacted.
* Meet specific risk-group requirements, for women at heterosexual risk, for men at heterosexual risk, and for injection drug users.

Exclusion Criteria

Participants will not be eligible for this study if they:

* Have any mental disorders that would cause a problem with the informed consent or study participation.
* Have any condition that, in the opinion of the doctor, would interfere with the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000
Dates: Start 2002-04; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ryder, Study Chair
Locations (3):
- China (2):
  - Guangxi Ctrs. for Disease Control & Prevention and for HIV/AIDS Prevention & Control CRS, Nanning, Guangxi
  - Xinjiang Uygar Autonomous Region Ctr. for Disease Control & Prevention, HPTN Project Office, Ürümqi, Xinjiang
- St. Petersburg Univ. Biomedical Ctr., Saint Petersburg, Russia